CLINICAL TRIAL: NCT04612621
Title: MILESTONE-CD -A Prospective Multiomic Inception Real -Life Study To Evaluate Predictors of Disease Outcomes & respoNse to Biologic Treatment in Crohn's Disease
Acronym: MILESTONE-CD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHEBA-20-7346-UK-CTIL
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Crohn Disease of Intestine

STUDY DESIGN:
Intervention Model Description: All enrolled patients will undergo similar interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: combination of diagnostic tests — capsule endoscopy, MRE , intestinal ultrasound, fecal microbiota, blood and serum biomarkers as described

SUMMARY:
Crohn's' disease (CD) is a lifelong-chronic inflammatory condition of the digestive tract. CD frequently manifests during the 2nd or 3rd decade; prolonged disease duration frequently results in major structural complications such as strictures and fistulae, leading to surgery for control of complications in at least 30% of the patients. The course of disease is extremely diverse, ranging from a very mild disease to a devastating and incapacitating course. The burden of inflammatory bowel disease is growing each disease, reaching 400 billion USD for lifetime in US. In Israel, there are currently over 50000 IBD patients, with one of the highest incidences in the word, multiple treatment modalities and medications are available for Crohn's disease, however the efficacy is limited and the costs- very high. Furthermore, long-term exposure to some of the therapeutic agents poses an increased risk of infections and cancer.

Some of the major challenges in IBD include prediction of disease course (some patients will require early and aggressive treatment while others may just need observation and follow-up), and treatment personalization (right drug for the right patient at the right time). Unfortunately, individualized predictors of disease course and response to treatment are currently very limited. Some clues can be derived from imaging and endoscopy data, transcriptomics, genomic and microbiome, however those are still very premature and impractical. Moreover, large-scale studies with sophisticated predictive models that incorporate multilayered and multilayered clinical and omic data are severely lacking.

DETAILED DESCRIPTION:
Goal:

Create comprehensive patient-multiomic profile (PRO-Visualosome-microbiome-transcriptome-pharmacokineticome) to develop algorithm-based personalized IBD therapy

Design Prospective observational cohort study.

Study aim To detect predictors of response to biologics using a layered multiomic approach

Cohort size Up to 140 patients in 2 years

Study duration -Patients will be followed up to 2 years (possible extension) or until treatment discontinuation or intestinal surgery

Study procedures All study procedures will be performed for the purpose of the study

Baseline

Disease activity using Harvey Bradshaw score at all timepoints and visits

* baseline PROS -PROMIS10/SIBDQ/IBD control/PRO2 using DATOS app
* colonoscopy with Intestinal biopsies
* Blood for transcriptomics
* Blood/serum for serum and cellular markers
* Stool for microbiome/metabolomics (if colonoscopy done- a rectal swab during colonoscopy will be performed)
* Pillcam CD following patency capsule - if failed patients still will be included and continue follow- up without capsule endoscopy
* MRE
* IUS
* Fecal calprotectin home kit with CALPROSMART
* Basic chemistry
* Joint US (if joint symptoms) Repeated assessment -every month
* PROMIS10/SIBDQ/IBD control/-via DATOS app (during the first 14-16 weeks- PRO2 will be evaluated weekly) Continuous monitoring (mobile device via DATOS app)

First follow-up visit (12-14 weeks)

* Calprotectin
* Microbiome
* Blood for transcriptomics
* Blood/serum for serum and cellular markers, drug levels, CRP

Every 3 months

- Home calprotectin (Calprosmart) +microbiome

Every 6 months

* Clinic visit
* Pillcam CD
* IUS
* Blood for transcriptomics
* Blood/serum for serum and cellular markers, drug levels, CRP
* Calprotectin (home +ELISA) + microbiome

Upon failure (need to switch medication -defined by treating physician) or end of study

* Clinic visit
* Calprotectin *Home +ELISA)
* Microbiome
* Serum for transriptomics, metabolomics
* Blood/serum for serum and cellular markers, drug levels, CRP
* Repeat Pillcam CD (if not done within 6 months)
* Repeat IUS +thermal imaging (if not done within 6 months)
* MRE

  * Drug levels will be done at every infusion for IV drugs and every 6 months for SC biologics and at the end of induction (week 8-16)

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease
* Start of first-line biological therapy

Exclusion Criteria:

* Previous biologic therapy
* Previous surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
failure of first biologic | 2 years
  cessation or switch of first biologic as per decision of the treating physician (documentation of change of therapy from the first biologic for any reason)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No